CLINICAL TRIAL: NCT02450760
Title: Connected Health Blood Pressure Monitoring In Stroke and TIA Patients
Acronym: CHAMPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 821743
Record Dates: First submitted 2015-05-18; First posted 2015-05-21 (Estimated); Results first posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2021-12

CONDITIONS: Stroke; Ischemic Attack, Transient
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): Subjects will take their blood pressure twice daily using the provided Withings blood pressure cuff. If subjects miss blood pressure readings, they will receive automated alerts reminding them to take their blood pressure. Subjects will also receive weekly emails with their blood pressure data for the week.
  Interventions: Other: Social incentive
- Social Incentive (Other): Subjects will take their blood pressure twice daily using the provided Withings blood pressure cuff. Subjects in this arm will also identify a social supporter who may help subjects adhere to daily blood pressure readings. If the subject misses blood pressure readings, they will receive automated alerts reminding them to take their blood pressure. The identified social supporter will also receive these alerts, with the expectation that the social supporter will remind the subject to take their blood pressure. Both the subject and the social supporter will also receive weekly emails with their blood pressure data for the week.
  Interventions: Other: Social incentive

INTERVENTIONS:
Other: Social incentive — Quantify adherence to 90 days of home blood pressure monitoring and to determine if a social incentive improves adherence

SUMMARY:
The goal of this pilot project is to assess adherence with home blood pressure monitoring in hypertensive patients with a history of cerebral infarction and to determine if a social incentive improves adherence with monitoring. Enrolled subjects will all have a history of cerebral infarction and uncontrolled blood pressure, defined by SBP>140 or DBP>90 mm Hg at the time of enrollment. To be eligible subjects will also be required to own a smart phone (iOS or Android operating system). After enrollment, patients will be given a home blood pressure cuff with instructions to monitor their BP twice daily for 90 days. Subjects will be randomly assigned to a social incentive program, in which a social supporter receives updates via email and/or text message on the subject's adherence with BP monitoring and their average blood pressure. This study will provide important pilot data which will inform the design of future studies utilizing connected health and automated systems to improve home blood pressure monitoring and blood pressure control in patients with a history of stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adult, age ≥ 18 years
* History of ischemic stroke or high risk TIA (defined by ABCD2 ≥ 4)between 2 weeks and 12 months prior to enrollment
* Hypertensive at time of enrollment, defined by SBP>140 mm Hg or DBP >90 mm Hg at the time of study screening
* Must own a smart phone capable of interacting with the connected blood pressure cuff (Apple iPhone 3GS or higher; Android 4.0 or higher with Bluetooth connectivity)
* Willingness and ability to sign informed consent by patient

Exclusion Criteria:

* Moderate or severe disability, defined by modified Rankin Scale ≥ 3.
* Expected residence in a rehabilitation hospital, nursing facility or assisted living community during the study period.
* Upper arm circumference <9 inches or >17 inches
* Inability to monitor BP in both of the upper arms (i.e. history of bilateral radical mastectomy, bilateral severe subclavian stenosis, or bilateral arterial venous fistulas for dialysis).
* Blood pressure discrepancy between arms of >10 mm Hg.
* Inability to follow-up at 90 days and return BP monitor
* Active participation in another clinical trial
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2021-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mullen, M.D, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Social Incentive
Started | 15 | 18
Completed | 15 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Social Incentive | Total
Number analyzed (Participants) | 15 | 18 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (9.3) | 59.4 (8.6) | 58.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 7 | 16
  White | 6 | 10 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 18 | 33

OUTCOME MEASURES:

1. Primary Outcome: Adherence With Home Blood Pressure Monitoring, Defined by the Proportion of Home Blood Pressure Recordings Successfully Completed
Description: Percentage of requested blood pressure measurements completed. Note that subjects were enrolled for 90 +/- 7 days, and so this calculation was completed at day 83, rather than day 90.
Time Frame: 90 Days
Population: All enrolled subjects
Measure: Median (Inter-Quartile Range); unit: percentage of requested BP measurements
Arm/Group | Control | Social Incentive
Number analyzed (Participants) | 15 | 18
percentage of requested BP measurements | 40 [16 to 73] | 60 [31 to 91]
Statistical Analysis 1: Comparison: Control vs Social Incentive; Test type: Superiority; p = 0.29, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Systolic Blood Pressure Over Study Period
Description: Difference in systolic blood pressure from the first 7 days of measurement to the last 7 days of measurement for each subject
Time Frame: 90 days
Population: Enrolled subjects
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control | Social Incentive
Number analyzed (Participants) | 15 | 18
mm Hg | 3.1 (14.0) | 2.7 (14.6)
Statistical Analysis 1: Comparison: Control vs Social Incentive; Test type: Superiority; p = 0.95, t-test, 2 sided

3. Secondary Outcome: Number of Physician Visits
Time Frame: 90 days
Population: Subjects who completed day 90 interview
Measure: Median (Inter-Quartile Range); unit: physician visits
Arm/Group | Control | Social Incentive
Number analyzed (Participants) | 8 | 13
physician visits | 2 [2 to 3.5] | 3 [2 to 4]

4. Secondary Outcome: Number of Emergency Department Visits
Time Frame: 90 days
Population: Subjects who completed day 90 interview
Measure: Median (Inter-Quartile Range); unit: Number of ED visits
Arm/Group | Control | Social Incentive
Number analyzed (Participants) | 8 | 13
Number of ED visits | 0 [0 to 0] | 1 [1 to 2]

5. Secondary Outcome: Number of Changes in Antihypertensive Medications (Dose Adjustment or Addition of a New Agent)
Time Frame: 90 days
Population: subjects completing day 90 interview
Measure: Median (Inter-Quartile Range); unit: Number of changes to BP medications
Arm/Group | Control | Social Incentive
Number analyzed (Participants) | 8 | 13
Number of changes to BP medications | 0 [0 to 1] | 0 [0 to 1]

6. Secondary Outcome: Number of Participates That Perceived the Blood Pressure Monitoring Device to be Easy to Use
Description: Number of patients who felt that device was easy or very easy to use
Time Frame: 90 days
Population: 24 subjects completed 90 day survey
Measure: Count of Participants; unit: Participants
Groups:
- Social Support: Social support intervention group
- Control: Control group
Arm/Group | Social Support | Control
Number analyzed (Participants) | 14 | 10
Participants | 9 | 9
Statistical Analysis 1: Comparison: Social Support vs Control; Test type: Superiority; p = 0.15, Chi-squared

7. Secondary Outcome: Number of Patients That Perceived Blood Pressure Monitoring to be Useful
Description: Number of participants who felt that BP monitoring was useful or very useful
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Groups:
- Social Support: Social support intervention arm
- Control: Control Arm
Arm/Group | Social Support | Control
Number analyzed (Participants) | 14 | 10
Participants | 4 | 3
Statistical Analysis 1: Comparison: Social Support vs Control; Test type: Superiority; p = 0.83, Chi-squared

8. Secondary Outcome: Number of Patients Who Felt They Had Well-controlled Blood Pressure
Description: Patients perception of whether or not BP was well controlled
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Groups:
- Social Support: Social Support Arm
Arm/Group | Social Support | Control
Number analyzed (Participants) | 14 | 10
Participants | 10 | 9
Statistical Analysis 1: Comparison: Social Support vs Control; Test type: Superiority; p = 0.26, Chi-squared

ADVERSE EVENTS:
Time Frame: 90 days
Description: Does not differ
Arm/Group | Control | Social Incentive
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/18
Other Adverse Events (participants affected / at risk) | 0/15 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT02450760/Prot_SAP_000.pdf